CLINICAL TRIAL: NCT05449964
Title: Comparative Evaluation of Outcomes of Single Sitting Scaling and Root Planing (SRP) vs Supra-gingival Scaling Followed by Sub-gingival Scaling and Root Planing After One Week: a Split-mouth Randomised Controlled Clinical Trial
Brief Title: Single Sitting SRP vs Supra-gingival Scaling Followed by Sub-gingival SRP After One Week
Acronym: SRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AANCHAL SAHNI PERIO
Record Dates: First submitted 2022-05-28; First posted 2022-07-08 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-07

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEST GROUP (Experimental): INTERVENTION: Scaling and root planning (SRP) of two contra-lateral quadrants (randomly allocated) in single sitting with ultrasonic scaler, hand scalers and curettes under local anaesthesia.
  Interventions: Procedure: SCALING AND ROOT PLANING (SRP)in single sitting
- CONTROL GROUP (Active Comparator): INTERVENTION: Supra-gingival scaling followed by sub-gingival scaling and root planing of two contra-lateral quadrants (randomly allocated) in two sittings with ultrasonic scaler, hand scalers and curettes under local anaesthesia.
  Interventions: Procedure: SCALING AND ROOT PLANING (SRP)in two sittings

INTERVENTIONS:
Procedure: SCALING AND ROOT PLANING (SRP)in single sitting — SCALING AND ROOT PLANING (SRP) IS THE PRIMARY COURSE OF NON-SURGICAL PERIODONTAL TREATMENT THAT INVOLVES REMOVAL OF SUPRA-GINGIVAL AND SUB-GINGIVAL BIOFILM AND CALCULUS FOLLOWED BY THOROUGH ROOT PLANING.
  Arms: TEST GROUP
Procedure: SCALING AND ROOT PLANING (SRP)in two sittings — SCALING AND ROOT PLANING (SRP) IS THE PRIMARY COURSE OF NON-SURGICAL PERIODONTAL TREATMENT THAT INVOLVES REMOVAL OF SUPRA-GINGIVAL AND SUB-GINGIVAL BIOFILM AND CALCULUS FOLLOWED BY THOROUGH ROOT PLANING.
  Arms: CONTROL GROUP

SUMMARY:
The primary course of periodontal treatment is non-surgical periodontal therapy followed by surgical therapy, if required, with an aim to arrest ongoing inflammatory periodontal destruction along with reconstruction of lost apparatus if possible. There is no protocol established for completing scaling and root planing (SRP) in patients with generalized advanced periodontitis. In some cases SRP is completed in single sitting whereas in other cases supragingival scaling is followed by subgingival SRP in the next appointment. It is hypothesized that presence of reparative components near the base of the pocket could result in better treatment outcomes after scaling and root planning done in single sitting when compared to supragingival scaling followed by sub-gingival scaling and root planning after one week.

DETAILED DESCRIPTION:
The aim of this randomized controlled clinical trial is to clinically compare the outcomes of scaling and root planing (SRP) completed in single sitting vs supragingival scaling followed by subgingival scaling and root planing after one week in Stage II and Stage III generalised periodontitis patients.

OBJECTIVES:

1. To assess the improvement in clinical parameters viz. bleeding on pocket probing (BOPP), pocket probing depth (PPD), clinical attachment level (CAL), plaque index (PI), gingival index (GI), bleeding on marginal probing (BOMP), gingival marginal position (GMP) and gingival recession (GR) by single sitting scaling and root planning versus supragingival scaling followed by subgingival scaling and root planing after one week in Stage II and Stage III generalised periodontitis patients.
2. To assess the correlation between availability of Vascular Endothelial Growth Factor (VEGF) at the base of the pocket and treatment outcomes.

SETTING: Department of Periodontology and Oral Implantology, PGIDS, Rohtak, Haryana.

STUDY DESIGN: Split-mouth Randomized controlled clinical trial.

TIME FRAME: 12 months

POPULATION: Systemically healthy patients with Stage II and Stage III Generalised Periodontitis with more than 20 teeth present.

SAMPLE SIZE: To be able to detect a clinically meaningful difference of 1mm and 10% improvement in PPD and BOPP respectively between groups, assuming an effect size of 0.85 with a power of 80% and 5% level of significance, a minimum sample size of 22 patients are needed in each group. Accounting for a 20% drop out rate, 27 patients are needed in each group.

METHODOLOGY: Patients with stage II and III generalised periodontitis will be recruited from the outpatient Department of Periodontology, PGIDS, Rohtak. Patients fulfilling the eligibility criteria will be enrolled in the study after obtaining an informed written consent. A split-mouth design will be chosen using two contra-lateral quadrants per group being randomly assigned into test (single sitting SRP) and control (supragingival scaling followed by subgingival scaling after a week) group for each patient using a chit-method.

ELIGIBILITY:
Inclusion Criteria:

•Systemically healthy patients with Stage II and Stage III Generalised Periodontitis with more than 20 teeth present.

Exclusion Criteria:

* Systemic illness known to affect the periodontium or outcome of periodontal therapy.
* Mobile teeth (Mobility no. 2 and 3 as per Miller Index)
* Patient taking medications such as NSAIDS, corticosteroids, statins or calcium channel blockers, which are known to interfere with periodontal wound healing.
* Pregnant or lactating women.
* History of use of tobacco.
* History of periodontal treatment in last 2 years.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change in bleeding on pocket probing (BOPP) | 6 MONTHS
  CHANGE IN BLEEDING ON POCKET PROBING FROM BASELINE TO 6 MONTHS
Chane in pocket probing depth (PPD) | 6 MONTHS
  CHANGE IN POCKET PROBING DEPTH FROM BASELINE TO 6 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: AANCHAL SAHNI, BDS, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES,ROHTAK
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahni A, Sharma RK, Tewari S, Gill PS, Arora R. Impact of supragingival scaling on the outcomes of subgingival instrumentation completed after 1 week: a split-mouth randomized clinical trial. Quintessence Int. 2023 Oct 19;54(9):724-733. doi: 10.3290/j.qi.b4168461. PMID 37334784